CLINICAL TRIAL: NCT03122392
Title: Pressure-Volume Measurements on the AMS 800TM Cuff
Acronym: AUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1703M09441
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Volume and Pressure Profiles in the AMS 800 cuff. The cuff is filled with deionized water and the amount of fluid in it decides the pressure it will apply while wrapped around the urethra. The pressure-volume profiles will be taken from 6 patients consented by the PI and these will be used for the secondary end point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- AMS 800 Artificial Urinary Sphincter (Experimental): The AMS 800™ Urinary Control System is an implantable, fluid-filled, solid silicone elastomer prosthesis used to treat urinary incontinence due to reduced outlet resistance (intrinsic sphincter deficiency) following prostate surgery. The AMS 800 Urinary Control System simulates normal sphincter function by opening and closing the urethra, under patient control. When the cuff is closed, urine stays in the bladder.
  When the patient wishes to void, he simply squeezes and releases the pump several times. This causes the fluid in the cuff to move into the pressure-regulating balloon . The cuff opens and urine passes through the urethra. The balloon then automatically re-pressurizes the cuff through the pump, within several minutes, the cuff again closes the urethra.
  The control pump, which in implanted in the scrotum, is also designed to allow the clinician or patient to deactivate and activate the system without additional surgery.
  Interventions: Device: AMS 800

INTERVENTIONS:
Device: AMS 800 — AMS 800 Artificial Urinary Sphincter

SUMMARY:
he idea of the experiment is to calculate the volume of fluid that is required to raise cuff pressure from 20 cmH2O to 120 cmH2O in the American Medical System's AMS 800 Artificial Urinary Sphincter (AUS).

DETAILED DESCRIPTION:
The current AMS 800 is not personalized to the patient's needs. Most men only need 20 cm H2O of urethral compression to remain dry when they are sedentary, yet need 120 cm H2O of urethral compression when they are active. The current device compromises with an in between pressure - as high as it can be without exceeding safety tolerance thresholds. As such many men still leak when they are active. In fact, this compromise is so central to the device that a new term has evolved to describe men's suboptimal level of continence after the AMS 800. We call it "social continence", meaning that they are dry enough to only have to wear 1-2 pads per day for protection.

The market is hungry for a device that can adapt to the patient's level of activity, reducing the pressure most of the day to protect the urethra and then briefly increasing the pressure when he is more active.

The experimental procedure is explained below and care will be taken to make sure the pressure sensor is sterile. The experiment involves minimal risk and will be conducted by the PI who has 10+ years of experience in AUS implantations.

The procedure for implanting the AMS 800 is mentioned in the Operating Manual attached with this protocol. The treatment procedure is linked with the experimental setup designed by the PI and the research student in the following manner:

1. Follow surgical preparation steps mentioned on pages 14-15 of the AMS 800 Operating Manual. Once the cuff sizer is used to determine the cuff length (usually 4.0cm or 4.5cm), move on to next step. For graphical representation, follow steps 1 to 9b on pages 18- 20 of the AMS 800 Operating Manual.
2. The AMS 800 cuff is filled with deionized water such that pressure is 20cmH2O. Follow steps on pages 13-14 of the AMS 800 Operating Manual for filling the cuff.
3. The AMS 800 cuff around the urethra has a kink-free tubing which goes into a female connector
4. The female connector connects to the male connector of the IV tubing
5. The IV tubing is connected to a T-Connector
6. One end of the T-Connector goes to the TruWave Pressure Transducer
7. Other end goes to a syringe
8. The system is pumped with deionized water and is therefore sterile.
9. Water is pumped into the cuff with the syringe and as the volume in the cuff increases, corresponding cuff pressure changes. This is done until we have a volume for a pressure reading of 120cmH2O on the pressure transducer.
10. Once the reading is obtained, the PI will flush out the excess water from the cuff, and fill it with an optimal volume as required by the treatment procedure which he has performed for over 10 years.
11. The treatment procedure will continue to follow the steps hereafter as has been designed for AUS placement.

For all other details including device description and post-operative care, refer to the AMS 800 operating Manual. All devices including the AMS 800 (PMA-P000053) and the Edward LifeSciences Pressure Transducer (501K- K142749) are FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 100 years of age who are to undergo AUS placement for treatment of stress urinary incontinence.

Exclusion Criteria:

* Under the age of 18 years old English non-speaking Unable to consent for themselves If a trans-corporal technique to AUS implantation is planned as this may affect the pressure measurements (<10% of the AUSs we implant are transcorporal).

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Pressure-Volume Measurements on the AMS 800TM Cuff | 6 months
  Measure volume and corresponding pressure in AMS 800TM occlusion Cuff

CONTACTS AND LOCATIONS:
Overall Officials: Sean Elliot, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No